CLINICAL TRIAL: NCT05053113
Title: A Peer-Based Approach to Enhance Physical Activity in Dyads of Inactive Women
Brief Title: Utilization of a Peer-Based Approach for the Promotion of Physical Activity in Inactive Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Heart, Lung, and Blood Institute should be included as a Collaborator. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020-0809; NCI-2020-13914 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0809 (Other: M D Anderson Cancer Center); R01HL155310 (NIH)
Record Dates: First submitted 2021-09-08; First posted 2021-09-22 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Obesity-Related Malignant Neoplasm
MeSH Terms: interventions — Fitness Trackers; Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (phone call, FitBit, newsletter, accelerometer) (Experimental): Participants receive phone calls over 30-45 minutes each from a health coach weekly during month 1, twice monthly during months 2-4, and monthly during months 5-6 for a total of 12 phone calls that focus on identifying needs, practicing autonomy supportive behaviors, and the development of a mutual support plan. Participants also engage in at least one physical activity per week with their partner and monitor their own and each other's activity using a FitBit. Participants also wear an accelerometer for a minimum of 10 hours a day for 7 days. Participants also receive an electronic newsletter twice monthly during months 1-3 and monthly during months 4-6 that provides educational physical activity-related information and tips for overcoming barriers to physical activity.
  Interventions: Device: Activity Monitor; Other: Educational Intervention; Other: Survey Administration; Behavioral: Telephone-Based Intervention
- Group 2A (phone call, FitBit, newsletter, accelerometer) (Active Comparator): Participants receive phone calls from a health coach as in Intervention I that focus on providing support for behavioral skills, including monitoring physical activity, goal-setting, and problem-solving to overcome barriers to physical activity. Participants utilize a FitBit to monitor their physical activity and receive electronic newsletters twice monthly during months 1-3 and monthly during months 4-6 that provides educational physical activity-related information and tips for overcoming barriers to physical activity. Participants also wear an accelerometer for a minimum of 10 hours a day for 7 days.
  Interventions: Device: Activity Monitor; Other: Educational Intervention; Other: Survey Administration; Behavioral: Telephone-Based Intervention
- Group 2B (FitBit, newsletter, accelerometer) (Active Comparator): Participants utilize a FitBit to monitor their physical activity and receive electronic newsletters twice monthly during months 1-3 and monthly during months 4-6 to share basic health education related to physical activity and provide support for engagement. Participants also wear an accelerometer for a minimum of 10 hours a day for 7 days.
  Interventions: Device: Activity Monitor; Other: Educational Intervention; Other: Survey Administration

INTERVENTIONS:
Device: Activity Monitor — Monitor physical activity with FitBit
  Other Names: Activity Tracker; Activity Tracker Device; Physical Activity Measuring Device
Device: Activity Monitor — Wear accelerometer
  Other Names: Activity Tracker; Activity Tracker Device; Physical Activity Measuring Device
Other: Educational Intervention — Receive educational newsletter
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Survey Administration — Ancillary studies
Behavioral: Telephone-Based Intervention — Receive phone call from health coach
  Arms: Group 1 (phone call, FitBit, newsletter, accelerometer); Group 2A (phone call, FitBit, newsletter, accelerometer)

SUMMARY:
This clinical trial tests the effect of a physical activity intervention that emphasizes support between partners in women who are not physically active. Decisions about and participation in physical activity often involve others in one's social circle, including family and friends. Social support for physical activity and having someone with whom to engage in physical activity may promote behavioral change and help increase moderate-intensity physical activity in inactive women.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine whether the dyadic behavioral intervention produces greater engagement of moderate-intensity objective physical activity (PA) compared with the individual behavioral intervention.

SECONDARY OBJECTIVES:

I. Determine the effects of the dyadic behavioral intervention on hypothesized intervention mechanisms (e.g., autonomous motivation, social support, autonomy support, self-efficacy), and the associations of those mechanisms with PA outcomes.

II. Determine the effects of the dyadic behavioral intervention on secondary outcomes (i.e., self-reported moderate-intensity PA, lower body strength, blood pressure, anthropometric measures, mean daily steps, sedentary time) compared with the individual behavioral intervention.

III. Determine whether the dyadic behavioral intervention produces greater engagement of moderate-intensity PA compared with the individual control.

OUTLINE: Participants are randomized to 1 of 2 groups.

GROUP 1 (DYADIC INTERVENTION): Participants receive phone calls over 30-45 minutes each from a health coach weekly during month 1, twice monthly during months 2-4, and monthly during months 5-6 for a total of 12 phone calls that focus on identifying needs, practicing autonomy supportive behaviors, and the development of a mutual support plan. Participants also engage in at least one physical activity per week with their partner and monitor their own and each other's activity using a FitBit. Participants also wear an accelerometer for a minimum of 10 hours a day for 7 days. Participants also receive an electronic newsletter twice monthly during months 1-3 and monthly during months 4-6 that provides educational physical activity-related information and tips for overcoming barriers to physical activity.

GROUP 2 (INDIVIDUAL CONDITION): Participants are assigned to one of 2 groups.

GROUP 2A (INDIVIDUAL INTERVENTION): Participants receive phone calls from a health coach as in Intervention I that focus on providing support for behavioral skills, including monitoring physical activity, goal-setting, and problem-solving to overcome barriers to physical activity. Participants utilize a FitBit to monitor their physical activity and receive electronic newsletters twice monthly during months 1-3 and monthly during months 4-6 that provides educational physical activity-related information and tips for overcoming barriers to physical activity. Participants also wear an accelerometer for a minimum of 10 hours a day for 7 days.

GROUP 2B (HEALTH EDUCATION CONTROL): Participants utilize a FitBit to monitor their physical activity and receive electronic newsletters twice monthly during months 1-3 and monthly during months 4-6 to share basic health education related to physical activity and provide support for engagement. Participants also wear an accelerometer for a minimum of 10 hours a day for 7 days.

At completion of study, patients are followed up at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as female
* Age 18-65 years
* Speak English or Spanish
* Physically able to engage in low-to-moderate PA as assessed by the PA Readiness Questionnaire (PAR-Q), or with medical clearance
* Insufficient self-reported moderate-to-vigorous PA (< 150 minutes/week)
* Able to enroll with one eligible adult female partner
* Valid home address in the greater Houston area
* Have a functioning smartphone and able and willing to send and receive text messages
* Willing to use the Fitbit app and device
* Blood pressure reading < 160/100 mm Hg, or with medical clearance

Exclusion Criteria:

* Pregnancy or considering pregnancy during the study period, self-reported
* Currently participating in a program or research study to promote physical activity or weight loss
* Plans to move outside the greater Houston area during the study period

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-07-27 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Change in objective minutes per week of moderate-intensity physical activity | Through study completion, an average of 1 year
  Will use a linear mixed model (LMM) analysis, which includes the intervention as a fixed effect predictor and a dyad-specific random intercept to account for the dependent nature of the nested design (in the dyadic intervention group) to assess if the dyadic intervention led to increased moderate-intensity physical activity, relative to the individual intervention. will also assess changes in physical activity across time (i.e., at 6 and 12 months after baseline) using longitudinal data, where both within-dyad and within-subject (repeated measures across time points) correlations will be accounted for. Relevant covariates (e.g., age, race/ethnicity, dyad relationship, education, household income and composition, employment status, neighborhood environmental characteristics) will be adjusted for in the analysis. Potential effect modifiers, e.g., depressive symptoms, perceived stress, neighborhood environmental characteristics, will be explored.

CONTACTS AND LOCATIONS:
Overall Officials: Larkin Strong, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson Cancer Center — http://www.mdanderson.org